CLINICAL TRIAL: NCT03009019
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Efficacy, Tolerability, and Safety Study of DFN-15 in Episodic Migraine With or Without Aura
Brief Title: Efficacy, Tolerability, and Safety of DFN-15
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Collaborators: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFN-15-CD-006
Record Dates: First submitted 2016-12-27; First posted 2017-01-04 (Estimated); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFN-15 Active (Experimental): DFN-15 Active
  Interventions: Drug: DFN-15 Active
- DFN-15 Placebo (Placebo Comparator): DFN-15 Placebo
  Interventions: Other: DFN-15 Placebo

INTERVENTIONS:
Drug: DFN-15 Active
  Other Names: Celecoxib Oral Solution
  Arms: DFN-15 Active
Other: DFN-15 Placebo
  Arms: DFN-15 Placebo

SUMMARY:
Efficacy, Tolerability, and Safety of DFN-15 in episodic migraine with or without aura, being conducted at multiple centers in the United States

ELIGIBILITY:
Inclusion Criteria:

1. A history of episodic migraine, who experience 2 to 8 migraine attacks per month for at least the past 12 months, with no more than 14 headache days per month, and with 48 hours of headache-free time between migraine attacks.
2. Patients who have migraine with or without aura with onset before age 50 years
3. Report usual migraine pain of 2 (moderate) or 3 (severe) on headache pain severity scale without treatment.
4. Subjects who are willing and able to:

   1. Evaluate and record pain, migraine symptoms, and study drug effectiveness information in real-time using a subject eDiary for the duration of the study;
   2. Record each instance of the use of study drug and rescue medication in real-time using a subject eDiary for the duration of the study;
   3. Comply with all other study procedures and scheduling requirements.

Exclusion Criteria:

1. Minors, even if they are in the specified study age range
2. Medication overuse:

   1. Opioids greater than or equal to 10 days during the 90 days prior to screening
   2. Combination medications (e.g., Fiorinal®) greater than or equal to 10 days during the 90 days prior to screening (applies only if includes opioid and/or barbiturate)
   3. Nonsteroidal Anti-inflammatory Drugs or other simple medications greater than 14 days a month during the 90 days prior to screening
   4. Triptans or ergots greater than or equal to 10 days a month during the 90 days prior to screening
3. Treated with onabotulinumtoxin A (Botox®) for migraine within 4 months prior to screening. (If treated for cosmetic reasons, subjects may be included).
4. Current treatment with antipsychotics or use of antipsychotics within 30 days prior to randomization.
5. Patients who have received treatment with an investigational drug or device within 30 days of randomization, or participated in a central nervous system clinical trial within 2 months prior to randomization
6. Patients with positive screening test for human immunodeficiency virus [HIV], positive hepatitis B surface antigen (HBsAg), or positive hepatitis C virus [HCV] antibody
7. Subjects who are employees or immediate relatives of the employees of the Sponsor, any of its affiliates or partners, or of the clinical research study site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2016-12; Primary Completion 2017-11 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Site 609, Birmingham, Alabama
  - Site 640, Mobile, Alabama
  - Site 622, Tucson, Arizona
  - Site 616, Hot Springs, Arkansas
  - Site 637, Huntington Beach, California
  - Site 615, Oakland, California
  - Site 646, San Diego, California
  - Site 619, San Francisco, California
  - Site 624, San Marcos, California
  - Site 631, Littleton, Colorado
  - Site 603, Miami, Florida
  - Site 641, Orange City, Florida
  - Site 629, Orlando, Florida
  - Site 601, West Palm Beach, Florida
  - Site 625, Decatur, Georgia
  - Site 630, Sandy Springs, Georgia
  - Site 642, Meridian, Idaho
  - Site 604, Blue Island, Illinois
  - Site 602, Louisville, Kentucky
  - Site 644, New Orleans, Louisiana
  - Site 610, New Orleans, Louisiana
  - Site 634, Ann Arbor, Michigan
  - Site 623, Edina, Minnesota
  - Site 638, City of Saint Peters, Missouri
  - Site 606, Missoula, Montana
  - Site 613, Omaha, Nebraska
  - Site 647, Lebanon, New Hampshire
  - Site 618, Nashua, New Hampshire
  - Site 636, Albuquerque, New Mexico
  - Site 645, Brooklyn, New York
  - Site 608, Rochester, New York
  - Site 620, High Point, North Carolina
  - Site 643, Mooresville, North Carolina
  - Site 626, Fargo, North Dakota
  - Site 628, Cleveland, Ohio
  - Site 614, Warwick, Rhode Island
  - Site 639, Mt. Pleasant, South Carolina
  - Site 612, Dakota Dunes, South Dakota
  - Site 627, Austin, Texas
  - Site 611, Dallas, Texas
  - Site 632, San Antonio, Texas
  - Site 621, Taylorsville, Utah
  - Site 635, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lipton RB, Munjal S, Tepper SJ, Iaconangelo C, Serrano D. A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Tolerability, and Safety of Celecoxib Oral Solution (ELYXYB) in Acute Treatment of Episodic Migraine with or without Aura. J Pain Res. 2021 Aug 19;14:2529-2542. doi: 10.2147/JPR.S322292. eCollection 2021. PMID 34447267
- See also: Publication of study results — https://pubmed.ncbi.nlm.nih.gov/34447267/

RESULTS

PARTICIPANT FLOW:
Groups:
- DFN-15: Subjects who received DFN-15 (active study drug)
- Placebo: Subjects who received placebo equivalent for DFN-15
Period: Double-blind Period 1 (DB1)
Arm/Group | DFN-15 | Placebo
Started (Randomized) | 316 (4 subjects included in the 'Started' & 'Not Completed' tallies were randomized but not dosed) | 315 (2 subjects included in the 'Started' & 'Not Completed' tallies were randomized but not dosed)
Completed (Completed DB1) | 280 | 264
Not Completed | 36 | 51
Period: Double-blind Period 2 (DB2)
Arm/Group | DFN-15 | Placebo
Started (Re-randomized for DB2) | 272 (4 subjects included in the 'Started' & 'Not Completed' tallies were randomized but not dosed) | 273 (1 subject included in the 'Started' & 'Not Completed' tallies was randomized but not dosed)
Completed (Completed DB2) | 251 | 253
Not Completed | 21 | 20

BASELINE CHARACTERISTICS:
Population: Safety Set 1 (for DB1)
Groups:
- DB1 Placebo: Subjects received placebo in the Double-blind period 1 (DB1)
- DB1 DFN-15: Subjects received DFN-15 in the Double-blind period 1 (DB1)
- Total: Total of all reporting groups
Arm/Group | DB1 Placebo | DB1 DFN-15 | Total
Number analyzed (Participants) | 283 | 289 | 572
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (12.99) | 41.4 (13.94) | 41.0 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 237 | 482
  Male | 38 | 52 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 40 | 81
  Not Hispanic or Latino | 241 | 248 | 489
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 63 | 64 | 127
  White | 209 | 214 | 423
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Are Pain-free at 2 Hours Postdose (First Treated Double-blind Treatment Period)
Description: The primary efficacy end point (for first treated DB1 attack only) were the percentage of subjects who were pain-free 2 hours postdose compared between DFN-15 and placebo (defined as a reduction from predose moderate [Grade 2] or severe [Grade 3] pain to none [Grade 0]
Time Frame: 2 hours postdose
Population: Full Analysis Set 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- DFN-15 Placebo (LOCF); DFN-15 Active (LOCF): last observation carried forward (LOCF)
- DFN-15 Placebo (OC); DFN-15 Active (OC): observed cases (OC)
Arm/Group | DFN-15 Placebo (LOCF) | DFN-15 Active (LOCF) | DFN-15 Placebo (OC) | DFN-15 Active (OC)
Number analyzed (Participants) | 267 | 280 | 256 | 275
percentage of subjects | 25.8 [20.7 to 31.5] | 32.9 [27.4 to 38.7] | 24.6 [19.5 to 30.4] | 32.4 [26.9 to 38.2]
Statistical Analysis 1: Comparison: DFN-15 Placebo (LOCF) vs DFN-15 Active (LOCF); Last Observation Carried Forward (LOCF); Test type: Superiority; p = 0.075, Fisher Exact; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.97 to 2.03]
Statistical Analysis 2: Comparison: DFN-15 Placebo (OC) vs DFN-15 Active (OC); Observed cases (OC); Test type: Superiority; p = 0.055, Fisher Exact; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.00 to 2.14]

2. Primary Outcome: Percentage of Subjects Who Are Free From Their MBS at 2 Hours Postdose
Description: Percentage of subjects who are free from their Most Bothersome Symptom (MBS) among nausea, photophobia, and phonophobia (first double-blind treatment period)
Time Frame: 2 hours postdose
Population: Full Analysis Set 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | DFN-15 Placebo (LOCF) | DFN-15 Active (LOCF) | DFN-15 Placebo (OC) | DFN-15 Active (OC)
Number analyzed (Participants) | 272 | 278 | 272 | 278
percentage of subjects | 45.0 [38.5 to 51.7] | 58.9 [52.4 to 65.2] | 44.4 [37.8 to 51.2] | 58.5 [51.9 to 64.8]
Statistical Analysis 1: Comparison: DFN-15 Placebo (LOCF) vs DFN-15 Active (LOCF); Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.22 to 2.52]
Statistical Analysis 2: Comparison: DFN-15 Placebo (OC) vs DFN-15 Active (OC); Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.22 to 2.55]

3. Secondary Outcome: The Number of Subjects With TEAEs After Study Drug Compared Between DFN-15 and Placebo
Description: For DB1: TEAE that started or worsening of a pre-existing condition on or after the first dose of study drug (DFN-15 or placebo) in to taking DB2 study drug, whichever occurs first.
  For DB2: TEAE that started or worsened on or after the first dose of study drug in DB2 up to 5 days after the date of the last dose of study drug in DB2.
Time Frame: Per protocol, the maximum dosing timeframe for DB2 was 10 weeks; therefore, the maximum AE collection window was 11 weeks total.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo DB1: Subjects with treatment-emergent adverse events (TEAEs) following placebo in the 1st double-blind treatment phase (DB1)
- DFN-15 DB1: Subjects with treatment-emergent adverse events (TEAEs) following DFN-15 in the 1st double-blind treatment phase (DB1)
- Placebo DB2: Subjects with treatment-emergent adverse events (TEAEs) following placebo in the 2nd double-blind treatment phase (DB2)
- DFN-15 DB2: Subjects with treatment-emergent adverse events (TEAEs) following DFN-15 in the 2nd double-blind treatment phase (DB2)
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 283 | 289 | 254 | 251
Participants | 28 | 31 | 26 | 21

4. Secondary Outcome: Freedom From Nausea, Photophobia, and Phonophobia Postdose (DB1 and DB2)
Description: The percentage of subjects who were free from nausea, photophobia, and phonophobia at 15, 30, and 45 minutes and 1, 1.5, 2, 4, and 24 hours postdose compared between DFN-15 and placebo
Time Frame: 15 minutes to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Placebo DB1 Nausea; DFN-15 DB1 Nausea; Placebo DB2 Nausea; DFN-15 DB2 Nausea: Subjects reporting nausea at time 0
- Placebo DB1 Photophobia; DFN-15 DB1 Photophobia; Placebo DB2 Photophobia; DFN-15 DB2 Photophobia: Subjects reporting photophobia at time 0
- Placebo DB1 Phonophobia; DFN-15 DB1 Phonophobia; Placebo DB2 Phonophobia; DFN-15 DB2 Phonophobia: Subjects reporting phonophobia at time 0
Arm/Group | Placebo DB1 Nausea | DFN-15 DB1 Nausea | Placebo DB1 Photophobia | DFN-15 DB1 Photophobia | Placebo DB1 Phonophobia | DFN-15 DB1 Phonophobia | Placebo DB2 Nausea | DFN-15 DB2 Nausea | Placebo DB2 Photophobia | DFN-15 DB2 Photophobia | Placebo DB2 Phonophobia | DFN-15 DB2 Phonophobia
Number analyzed (Participants) | 147 | 154 | 242 | 245 | 206 | 198 | 109 | 120 | 203 | 208 | 170 | 167
percentage of subjects
  15 minutes postdose | 20.3 [13.7 to 28.3] | 14.3 [8.8 to 21.4] | 6.2 [3.3 to 10.3] | 9.0 [5.5 to 13.6] | 11.1 [6.9 to 16.6] | 15.5 [10.5 to 21.8] | 10.4 [5.1 to 18.3] | 16.2 [9.7 to 24.7] | 3.3 [1.2 to 7.1] | 10.4 [6.4 to 15.8] | 8.7 [4.7 to 14.4] | 13.2 [8.1 to 19.8]
  30 minutes postdose | 35.3 [27.3 to 43.9] | 32.4 [25.0 to 40.6] | 14.7 [10.3 to 20.0] | 15.9 [11.4 to 21.2] | 16.8 [11.8 to 22.8] | 24.5 [18.5 to 31.3] | 27.5 [19.1 to 37.2] | 27.2 [19.3 to 36.3] | 15.0 [10.3 to 20.9] | 21.2 [15.7 to 27.6] | 19.5 [13.6 to 26.5] | 25.9 [19.3 to 33.5]
  45 minutes postdose | 40.3 [32.1 to 48.9] | 44.4 [36.3 to 52.7] | 22.8 [17.5 to 28.8] | 25.2 [19.8 to 31.2] | 29.4 [23.1 to 36.3] | 33.9 [27.2 to 41.0] | 40.4 [31.2 to 50.9] | 44.0 [34.8 to 53.5] | 25.3 [19.3 to 32.0] | 30.2 [23.9 to 37.0] | 29.2 [22.3 to 36.9] | 36.9 [29.4 to 44.9]
  1 hour postdose | 45.8 [37.4 to 54.3] | 55.9 [47.6 to 64.0] | 25.9 [20.4 to 32.0] | 32.0 [26.1 to 38.2] | 32.5 [26.0 to 39.5] | 39.5 [32.6 to 46.7] | 55.1 [45.2 to 65.8] | 56.9 [47.4 to 66.1] | 30.8 [24.5 to 37.7] | 37.2 [30.5 to 44.3] | 38.2 [30.7 to 46.1] | 48.1 [40.2 to 56.2]
  1.5 hours postdose | 53.5 [45.0 to 61.9] | 58.8 [50.6 to 66.7] | 35.6 [29.5 to 42.1] | 46.3 [39.9 to 52.8] | 40.9 [34.0 to 48.1] | 52.0 [44.8 to 59.2] | 58.9 [49.0 to 68.3] | 62.9 [53.5 to 71.7] | 42.2 [35.3 to 49.4] | 48.2 [41.1 to 55.4] | 52.4 [44.5 to 60.2] | 55.6 [47.6 to 63.5]
  2 hours postdose | 60.4 [51.9 to 68.5] | 66.7 [58.6 to 74.1] | 42.9 [36.5 to 49.4] | 58.0 [51.5 to 64.3] | 47.0 [40.0 to 54.2] | 59.2 [52.0 to 66.1] | 68.5 [58.9 to 77.1] | 72.9 [63.9 to 80.7] | 50.3 [43.1 to 57.4] | 53.7 [46.6 to 60.7] | 53.9 [46.0 to 61.6] | 61.3 [53.4 to 68.9]
  4 hours postdose | 74.0 [66.1 to 80.9] | 83.0 [76.1 to 88.6] | 57.5 [51.0 to 63.8] | 70.5 [64.3 to 76.1] | 65.2 [58.2 to 71.7] | 68.5 [61.5 to 74.9] | 73.1 [63.8 to 81.2] | 84.0 [76.2 to 90.1] | 61.0 [53.9 to 67.8] | 73.7 [67.1 to 79.5] | 69.5 [61.9 to 76.3] | 75.8 [65.5 to 82.1]
  24 hours postdose | 89.1 [82.9 to 93.6] | 89.6 [83.7 to 93.9] | 83.9 [78.6 to 88.3] | 86.5 [81.6 to 90.5] | 82.5 [76.6 to 87.4] | 88.9 [83.7 to 92.9] | 90.8 [83.8 to 95.5] | 93.3 [87.3 to 97.1] | 85.7 [80.1 to 90.2] | 90.4 [85.5 to 94.0] | 87.6 [81.7 to 92.2] | 89.2 [83.5 to 93.5]

5. Secondary Outcome: Time to Headache Pain Relief Postdose (DB1 and DB2)
Description: The time to headache pain relief was defined as the time in minutes from when a subject took study drug until the time pain relief was indicated by the subject in the eDiary within 2 hours postdose.
Time Frame: 2 hours postdose
Measure: Mean (95% Confidence Interval); unit: time (hours)
Groups:
- Placebo DB1: Placebo received in DB1
- DFN-15 DB1: DFN-15 received in DB1
- Placebo DB2: Placebo received in DB2
- DFN-15 DB2: DFN-15 received in DB2
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 44 | 34 | 29 | 29
time (hours) | NA [NA to NA] — Due to the small number of subjects who completed this assessment, the median time to headache pain relief was non-evaluable from the Kaplan-Meier survival estimation. | NA [NA to NA] — Due to the small number of subjects who completed this assessment, the median time to headache pain relief was non-evaluable from the Kaplan-Meier survival estimation. | NA [NA to NA] — Due to the small number of subjects who completed this assessment, the median time to headache pain relief was non-evaluable from the Kaplan-Meier survival estimation. | NA [NA to NA] — Due to the small number of subjects who completed this assessment, the median time to headache pain relief was non-evaluable from the Kaplan-Meier survival estimation.

6. Secondary Outcome: Time to Headache Pain Freedom Postdose (DB1 and DB2)
Description: The time to headache pain freedom was defined as the time in minutes from when a subject took study drug until the time pain freedom was indicated by the subject in the eDiary within 2 hours postdose.
Time Frame: 2 hours postdose
Measure: Median (95% Confidence Interval); unit: time (minutes)
Groups:
- Placebo DB1: Placebo received during DB1
- DFN-15 DB1: DFN-15 received during DB1
- Placebo DB2: Placebo received during DB2
- DFN-15 DB2: DFN-15 received during DB2
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 26 | 24 | 14 | 24
time (minutes) | NA [NA to NA] — Due to the small number of subjects who completed this assessment, time to headache pain freedom was non-evaluable from the Kaplan-Meier survival estimation | NA [NA to NA] — Due to the small number of subjects who completed this assessment, time to headache pain freedom was non-evaluable from the Kaplan-Meier survival estimation | NA [NA to NA] — Due to the small number of subjects who completed this assessment, time to headache pain freedom was non-evaluable from the Kaplan-Meier survival estimation | NA [NA to NA] — Due to the small number of subjects who completed this assessment, time to headache pain freedom was non-evaluable from the Kaplan-Meier survival estimation

7. Secondary Outcome: Headache Pain Relief Postdose (DB1 and DB2)
Description: Headache pain relief was defined for DB1 as a reduction from moderate or severe pain before dosing to mild or none postdose, and for DB2 as moderate or severe pain before dosing reduced to mild or none postdose, or mild pain before dosing reduced to none postdose. Data are reported by percentage reporting headache pain relief over time postdose.
Time Frame: 15 minutes to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Placebo DB1: Subjects received placebo in the 1st randomized double blind phase (DB1)
- DFN-15 DB1: Subjects received DFN-15 in the 1st randomized double blind phase (DB1)
- Placebo DB2: Subjects received placebo in the 2nd randomized double blind phase (DB2)
- DFN-15 DB2: Subjects received DFN-15 in the 2nd randomized double blind phase (DB2)
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
percentage of subjects
  15 minutes postdose | 12.6 [8.6 to 17.4] | 12.6 [8.7 to 17.3] | 7.9 [4.7 to 12.3] | 15.0 [10.5 to 20.4]
  30 minutes postdose | 22.4 [17.5 to 28.1] | 25.3 [20.2 to 30.9] | 23.0 [17.8 to 29.0] | 28.0 [22.3 to 34.3]
  45 minutes postdose | 35.0 [29.2 to 41.2] | 40.0 [34.2 to 46.1] | 35.3 [29.2 to 41.9] | 40.0 [33.7 to 46.6]
  1 hour postdose | 39.8 [33.9 to 46.1] | 49.6 [43.6 to 55.7] | 41.9 [35.6 to 48.5] | 52.8 [46.2 to 59.3]
  1.5 hours postdose | 49.6 [43.4 to 55.8] | 58.8 [52.8 to 64.6] | 51.9 [45.3 to 58.4] | 62.7 [56.2 to 68.9]
  2 hours postdose | 56.9 [50.8 to 62.9] | 68.6 [62.8 to 74.0] | 58.6 [52.0 to 64.9] | 69.6 [63.3 to 75.3]
  4 hours postdose | 73.8 [68.1 to 78.9] | 82.9 [78.0 to 87.1] | 74.6 [68.6 to 80.0] | 84.7 [79.5 to 89.0]
  24 hours postdose | 92.7 [89.0 to 95.5] | 94.3 [90.9 to 96.7] | 88.2 [83.4 to 91.9] | 95.1 [91.6 to 97.4]

8. Secondary Outcome: Headache Pain Freedom Postdose (DB1 and DB2)
Description: The percentage of subjects who were pain-free at 15, 30, and 45 minutes and 1, 1.5, 2 (DB2 period), 4, and 24 hours postdose compared between DFN-15 and placebo
Time Frame: 15 minutes to 24 hours postdose
Population: data for 2 hours postdose were not collected for DB1 per protocol
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
percentage of subjects
  15 minutes postdose | 2.9 [1.2 to 5.9] | 1.2 [0.3 to 3.5] | 0.5 [0.0 to 2.6] | 2.8 [1.0 to 6.0]
  30 minutes postdose | 5.5 [3.0 to 9.1] | 3.7 [1.8 to 6.7] | 1.7 [0.5 to 4.4] | 8.6 [5.3 to 13.0]
  45 minutes postdose | 9.7 [6.4 to 14.0] | 9.5 [6.3 to 13.5] | 7.3 [4.3 to 11.5] | 11.9 [8.1 to 16.8]
  1 hour postdose | 12.6 [8.9 to 17.3] | 18.0 [13.7 to 23.0] | 11.9 [8.0 to 16.7] | 18.7 [13.9 to 24.3]
  1.5 hours postdose | 19.8 [15.2 to 25.2] | 24.7 [19.8 to 30.2] | 20.7 [15.7 to 26.4] | 27.1 [21.6 to 33.3]
  2 hours postdose: number analyzed (Participants) | 0 | 0 | 253 | 250
  2 hours postdose |  |  | 24.3 [19.0 to 30.2] | 36.7 [30.6 to 43.1]
  4 hours postdose | 40.2 [34.3 to 46.3] | 49.1 [43.1 to 55.1] | 46.7 [40.2 to 53.2] | 59.1 [52.6 to 65.3]
  24 hours postdose | 71.9 [66.2 to 77.1] | 79.4 [74.2 to 84.0] | 74.7 [68.8 to 80.0] | 85.3 [80.2 to 89.5]

9. Secondary Outcome: Absence of Screening MBS at Time Points Postdose (DB1 and DB2)
Description: The percentage of subjects with their Screening MBS (Most Bothersome Symptom) absent at 15, 30, and 45 minutes and 1, 1.5, 2 (DB2 period), 4, and 24 hours postdose compared between DFN-15 and placebo.
Time Frame: 15 minutes to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
percentage of subjects
  15 minutes postdose | 8.3 [4.9 to 12.9] | 10.4 [6.6 to 15.3] | 5.8 [2.8 to 10.5] | 9.6 [5.7 to 14.9]
  30 minutes postdose | 17.0 [12.2 to 22.6] | 18.2 [13.4 to 23.8] | 16.4 [11.3 to 22.6] | 21.5 [15.9 to 28.0]
  45 minutes postdose | 24.0 [18.5 to 30.2] | 29.1 [23.4 to 35.3] | 28.1 [21.8 to 35.2] | 31.1 [24.6 to 38.1]
  1 hour postdose | 27.6 [21.8 to 33.9] | 36.0 [29.9 to 42.4] | 32.3 [25.7 to 39.4] | 42.0 [34.9 to 49.3]
  1.5 hours postdose | 38.1 [31.7 to 44.7] | 48.8 [42.3 to 55.3] | 44.7 [37.5 to 52.1] | 51.8 [44.5 to 59.0]
  2 hours postdose | 45.0 [38.5 to 51.7] | 58.9 [52.4 to 65.2] | 51.3 [44.0 to 58.6] | 56.9 [49.7 to 64.0]
  4 hours postdose | 61.4 [54.8 to 67.7] | 70.1 [36.9 to 75.8] | 61.5 [54.2 to 68.4] | 75.6 [69.0 to 81.5]
  24 hours postdose | 83.8 [78.4 to 88.2] | 86.4 [81.4 to 90.4] | 86.7 [81.1 to 91.1] | 91.0 [86.1 to 94.6]

10. Secondary Outcome: Change in Functional Disability Score Postdose (DB1 and DB2)
Description: Change in functional disability score at 2, 4, and 24 hours postdose compared between DFN-15 and placebo. The values of the functional disability scale were: 0=no disability, able to function normally; 1=performance of daily activities mildly impaired, can still do everything but with difficulty; 2=performance of daily activities moderately impaired, unable to do some things; 3=performance of daily activities severely impaired, cannot do all or most things, bed rest may be necessary.
  A decrease in values indicates improvement from baseline.
Time Frame: 2 to 24 hours postdose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
units on a scale
  2 hours postdose | -0.7 (0.95) | -0.9 (0.89) | -0.6 (0.94) | -0.9 (0.91)
  4 hours postdose | -1.0 (1.06) | -1.2 (0.89) | -0.9 (0.97) | -1.2 (0.90)
  24 hours postdose | -1.7 (0.92) | -1.7 (0.78) | -1.5 (0.84) | -1.7 (0.82)

11. Secondary Outcome: Headache Pain Freedom Among Subjects With Cutaneous Allodynia (DB1 and DB2)
Description: The percentage of subjects who were pain-free at 2 and 4 hours postdose compared between DFN-15 and placebo, among those reporting cutaneous allodynia predose
Time Frame: 2 and 4 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
percentage of subjects
  2 hours postdose | 26.2 [16.0 to 38.5] | 26.2 [15.8 to 39.1] | 25.5 [14.3 to 39.6] | 39.5 [25.0 to 55.6]
  4 hours postdose | 37.9 [26.2 to 50.7] | 39.3 [27.1 to 52.7] | 43.1 [29.3 to 57.8] | 54.5 [38.8 to 69.6]

12. Secondary Outcome: Headache Pain Freedom Among BMI Category (DB1 and DB2)
Description: The percentage of subjects who were pain-free at 2 and 4 hours postdose whose BMI was < 30 kg/m2 vs. subjects whose BMI was ≥ 30 kg/m2, and whose BMI was < 25 kg/m2 vs. subjects whose BMI was ≥ 25 kg/m2
Time Frame: 2 and 4 hours postdose
Population: Subjects were stratified and data were evaluated by subject BMI, therefore the overall number analyzed differs from the participant numbers reported in the data table.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
percentage of subjects
  2 hours postdose (BMI<30): number analyzed (Participants) | 144 | 156 | 122 | 140
  2 hours postdose (BMI<30) | 22.9 [16.3 to 30.7] | 25.6 [19.0 to 33.2] | 22.1 [15.1 to 30.5] | 34.3 [26.5 to 42.8]
  4 hours postdose (BMI<30): number analyzed (Participants) | 147 | 156 | 122 | 140
  4 hours postdose (BMI<30) | 38.1 [30.2 to 46.5] | 43.6 [35.7 to 51.8] | 44.3 [35.3 to 53.5] | 55.0 [46.4 to 63.4]
  2 hours postdose (BMI>=30): number analyzed (Participants) | 123 | 124 | 117 | 100
  2 hours postdose (BMI>=30) | 29.3 [21.4 to 38.1] | 41.9 [33.1 to 51.1] | 26.5 [18.8 to 35.5] | 40.0 [30.3 to 50.3]
  4 hours postdose (BMI>=30): number analyzed (Participants) | 124 | 125 | 118 | 102
  4 hours postdose (BMI>=30) | 42.7 [33.9 to 51.9] | 56.0 [46.8 to 64.9] | 49.2 [39.8 to 58.5] | 64.7 [54.6 to 73.9]

13. Secondary Outcome: Headache Pain Recurrence Postdose (DB1 and DB2)
Description: The percentage of subjects who had pain recurrence between 2 to 24 hours (i.e., pain-free at 2 hours postdose, with pain [mild, moderate, or severe] reported at 24 hours postdose) compared between DFN-15 and placebo
Time Frame: 2 to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
percentage of subjects | 10.1 [4.2 to 19.8] | 7.6 [3.1 to 15.1] | 6.9 [1.9 to 16.7] | 4.5 [1.3 to 11.1]

14. Secondary Outcome: Sustained Headache Pain Relief Postdose (DB1 and DB2)
Description: The percentage of the population of subjects who reported headache pain relief between 2 and 24 hours postdose.
Time Frame: 2 to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
percentage of subjects | 39.8 [33.0 to 46.9] | 55.1 [48.4 to 61.7] | 44.3 [37.0 to 51.8] | 56.6 [49.1 to 63.9]

15. Secondary Outcome: Sustained Headache Pain Freedom Postdose (DB1 and DB2)
Description: The percentage of subjects who had sustained pain freedom at 2 to 24 hours postdose compared between DFN-15 and placebo in each DB period. Sustained pain freedom at 2 to 24 hours postdose is defined as pain-free at 2 hours postdose, with no use of rescue medication, and no recurrence of headache pain within 2 to 24 hours postdose
Time Frame: 2 to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
percentage of subjects | 18.9 [13.7 to 25.0] | 27.6 [21.8 to 33.9] | 20.0 [14.5 to 26.5] | 29.1 [22.6 to 36.3]

16. Secondary Outcome: Use of Rescue Medication Postdose (DB1 and DB2)
Description: The percentage of subjects who used rescue medication after 2 hours (2 to 24 hours) postdose compared between DFN-15 and placebo in each DB period
Time Frame: 2 to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
percentage of subjects | 28.5 [23.2 to 34.2] | 18.8 [14.4 to 23.9] | 22.9 [17.8 to 28.6] | 18.4 [13.7 to 23.8]

17. Secondary Outcome: Subject-Rated Treatment Satisfaction Postdose (DB1 and DB2)
Description: Subject-rated treatment overall satisfaction was based on a 7-point scale at 2 and 4 hours postdose during each DB treatment period. The difference between the subject-rated study drug treatment satisfaction score at 2 and 4 hours postdose and the baseline PPMQ-R (Patient Perception of Migraine Questionnaire) response for the same question were summarized by treatment group (global satisfaction item at baseline asked about the subject's usual migraine treatment). The possible values of the subject treatment satisfaction scale were: 1=very satisfied, 2=satisfied, 3=somewhat satisfied, 4=neither satisfied nor dissatisfied, 5=somewhat dissatisfied, 6=dissatisfied, 7=very dissatisfied.
  A decrease in values indicates improvement from baseline.
Time Frame: 2 and 4 hours postdose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
units on a scale
  Difference at 2 hours | 0.7 (2.49) | -0.1 (2.35) | 0.3 (2.45) | -0.1 (2.26)
  Difference at 4 hours | 0.7 (2.50) | -0.1 (2.36) | 0.4 (2.46) | -0.1 (2.29)

18. Secondary Outcome: Subject-Rated Treatment Satisfaction at 24 Hours Postdose - PPMQ-R (DB1 and DB2)
Description: Patient Perception of Migraine Questionnaire-Revised had 30 questions assessing subject's satisfaction with migraine medication, including 3 global items & 4 subscales (i.e., efficacy, function, ease of use, tolerability). A 5-point scale (1-Not At All to 5-Extremely) was used for tolerability subscale questions; a 7-point scale (1-Very Satisfied to 7-Very Dissatisfied) was used for all other subscales and global items. Total score was average of efficacy/function/ease of use subscale scores. Each subscale & total scores were transformed to range from 0-100, with higher scores indicating better satisfaction or tolerability. Total raw score/global items were not transformed. The total raw score could range from 17 (min) to 119 (max), with lower scores indicating better satisfaction. Change from baseline scores at 24-hour-postdose for each subscale score, global item score, total score, & total raw score were summarized by treatment group below.
Time Frame: 24 hours postdose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 253 | 250
units on a scale
  Total Score | -4.866 (32.6258) | 5.112 (30.638) | 0.491 (32.5487) | 6.691 (28.1563)
  Total Raw Score | 2.463 (12.7476) | -1.498 (12.0209) | 0.426 (12.8385) | -2.312 (11.0429)
  Efficacy | -9.591 (41.0822) | 3.016 (38.9173) | -3.261 (41.6631) | 6.044 (36.1736)
  Function | -3.812 (42.0995) | 8.554 (39.4248) | 2.559 (42.3773) | 10.708 (35.2324)
  Ease of Use | -1.197 (29.1309) | 3.766 (26.0805) | 2.174 (27.7924) | 3.360 (23.7033)
  Tolerability | 6.09 (14.850) | 6.98 (15.267) | 5.87 (14.115) | 7.62 (17.579)
  Medication effectiveness (Global Item) | 0.9 (2.80) | 0.1 (2.64) | 0.6 (2.65) | -0.1 (2.43)
  Side Effects (Global Item) | -0.5 (2.00) | -0.4 (1.88) | -0.2 (1.98) | -0.5 (2.00)
  Overall Satisfaction (Global Item) | 0.8 (2.74) | 0.1 (2.60) | 0.5 (2.65) | -0.1 (2.41)

ADVERSE EVENTS:
Time Frame: Per protocol, the maximum dosing timeframe for DB2 was 10 weeks; therefore, the maximum AE collection window was 11 weeks total.
Description: For DB1: TEAE that started or worsening of a pre-existing condition on or after the first dose of study drug (DFN-15 or placebo) in to taking DB2 study drug, whichever occurs first.
  For DB2: TEAE that started or worsened on or after the first dose of study drug in DB2 up to 5 days after the date of the last dose of study drug in DB2.
  Overall group includes all subjects who received at least one dose of study drug (DFN-15 or placebo) during DB1.
Groups:
- Placebo DB1: TEAEs that occurred following placebo dose during DB1
- DFN-15 DB1: TEAEs that occurred following DFN-15 dose during DB1
- Placebo DB2: TEAEs that occurred following placebo dose during DB2
- DFN-15 DB2: TEAEs that occurred following DFN-15 dose during DB2
- Overall: TEAEs that occurred following the first dose of placebo or DFN-15
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2 | Overall
All-Cause Mortality (participants affected / at risk) | 0/283 | 0/289 | 0/254 | 0/251 | 0/572
Serious Adverse Events (participants affected / at risk) | 2/283 | 1/289 | 0/254 | 1/251 | 4/572
Other Adverse Events (participants affected / at risk) | 5/283 | 4/289 | 3/254 | 4/251 | 13/572
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo DB1 (N=283) | DFN-15 DB1 (N=289) | Placebo DB2 (N=254) | DFN-15 DB2 (N=251) | Overall (N=572)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 1
Pulmonary embolism (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cystitis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo DB1 (N=283) | DFN-15 DB1 (N=289) | Placebo DB2 (N=254) | DFN-15 DB2 (N=251) | Overall (N=572)
Nausea (Gastrointestinal disorders) | 5 | 4 | 3 | 4 | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT03009019/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03009019/SAP_001.pdf